CLINICAL TRIAL: NCT07015827
Title: Effect of Locally Produced Mango Variety on Glycemic Index
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, Naseer Ahmed, Associate proffessor, Rehman Medical Institute - RMI
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GL/GI-NA_1V1
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Glycemic Index and Glycemic Load
Keywords: Glycemic index; posprandial glucose response; glycemic load
MeSH Terms: interventions — Mangifera indica extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (cross over) (Active Comparator): Participants will consume 50 grams of glucose solution. This serves as the reference food for calculating the glycemic index
  Interventions: Other: Mango (langra); Other: mango (chaunsa); Other: MANGO (SINDHRI)

INTERVENTIONS:
Other: Mango (langra) — Participants will consume mango variety A . The test food will provide 50 grams of available carbohydrates, and will be consumed after an overnight fast.
Other: mango (chaunsa) — Participants will consume mango variety B . The test food will provide 50 grams of available carbohydrates, and will be consumed after an overnight fast.
Other: MANGO (SINDHRI) — Participants will consume mango variety C . The test food will provide 50 grams of available carbohydrates, and will be consumed after an overnight fast.

SUMMARY:
This randomized trial aims to assess the glycemic index (GI) of locally available mango varieties in healthy adult participants, using glucose as the reference food. The study will evaluate the postprandial blood glucose response elicited by selected mango varieties and compare it to the response produced by a standard glucose . The objective is to determine whether certain mango varieties have a lower glycemic impact, which may be relevant for dietary planning and public health recommendations.

DETAILED DESCRIPTION:
This randomized trial aims to assess the glycemic index (GI) of locally available mango varieties in healthy adult participants, using glucose as the reference food. The study will evaluate the postprandial blood glucose response elicited by selected mango varieties and compare it to the response produced by a standard glucose . The objective is to determine whether certain mango varieties have a lower glycemic impact, which may be relevant for dietary planning and public health recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-diabetic adults
* Normal fasting blood glucose levels
* Willingness to provide informed consent

Exclusion Criteria:

Diagnosis of diabetes mellitus or impaired glucose tolerance

* Gastrointestinal, metabolic, or endocrine disorders
* Current use of medications affecting blood glucose
* Pregnant or lactating women
* Smoking or alcohol consumption

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Glycemic Index (GI) of Mango Varieties | 0 to 120 minutes after consumption of test food
  Glycemic index will be calculated for each mango variety by measuring the postprandial blood glucose response over 120 minutes and comparing the incremental area under the curve (iAUC) to that of a standard glucose reference.

SECONDARY OUTCOMES:
Peak Blood Glucose Level | 0 to 120 minutes after consumption
  Maximum capillary blood glucose concentration observed after consumption of each test food.

IPD SHARING:
Plan to Share IPD: Undecided